CLINICAL TRIAL: NCT03874988
Title: Building an Evidence Base for Weight Loss Strategies Among Those With Chronic SCI-The GLB-SCI+
Acronym: GLB-SCI+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 018-783
Record Dates: First submitted 2019-02-07; First posted 2019-03-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Obesity; Weight Loss; Diet Modification
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Portion-Controlled Meals (Experimental): Participants will receive prepackaged food, delivered biweekly to their home over the course of 13 weeks, with costs covered by the grant. Depending on their calorie goals, participants will drink and eat a mix of shakes and entrees each day, plus up to five fruits and vegetables. HMR entrees and shakes are formulated to provide recommended levels of macronutrients, vitamins, sodium, fat, cholesterol and fiber and fortified to meet at least 100% of the recommended daily allowance for essential vitamins and minerals.
  Interventions: Behavioral: Portion-Controlled Meals
- Enhanced Self-Monitoring (Experimental): Participants will be encouraged to self-monitor 4 specific behaviors daily: 1) measuring their food; 2) measuring their physical activity; 3) recording their food, drink, and physical activity; and 4) monitoring their weight. To achieve this aim, participants will attend a single group-based educational session at baseline during which they will be provided the self-monitoring equipment (scale and Garmin vivofit) and receive training about how to use the Lilypad scale and smartphone food tracking app.
  Interventions: Behavioral: Enhanced Self-Monitoring
- GLB-SCI (Experimental): The content and delivery format of the developed GLB SCI lifestyle intervention program is subject to change based on guidance of the SCI Consumer Group. Therefore, this section provides a general description of the GLB AIM (lifestyle intervention program adapted for impaired mobility). The content of the GLB AIM core meetings include a mix of in-person (4) and telephone (9) sessions. The initial meeting is conducted in person, with one in-person sessions delivered each month, and the intervening weeks delivered by telephone. To achieve weight loss, participants will be encouraged to follow daily calorie and fat gram goals to achieve a .5 to 1 pound weight loss over the 13 weeks. Participants will also be encouraged to gradually increase their physical activity to ultimately achieve 150 weekly minutes.
  Interventions: Behavioral: GLB-SCI
- GLB-SCI+ (Experimental): The final multicomponent GLB SCI+ will include combining specific intervention strategies identified from the previous 3 interventions as effective and usable. If all 3 strategies yield evidence in support of being included, the combined intervention would encompass (1) providing prepackaged foods for a specified period of time to facilitate greater initial weight loss, (2) encouraging enhanced self-monitoring of food, physical activity, and weight using devices and apps along with social support, and (3) delivering the further adapted GLB SCI in a group-based format to teach skills helpful in making lifestyle changes.
  Interventions: Behavioral: GLB-SCI+

INTERVENTIONS:
Behavioral: Portion-Controlled Meals — Participants will receive portion-controlled meals with the aim of encouraging weight loss and healthier eating.
  Arms: Portion-Controlled Meals
Behavioral: Enhanced Self-Monitoring — Participants will be encouraged to track their physical activity, food intake, and weight using technology that will be provided as part of the study.
  Arms: Enhanced Self-Monitoring
Behavioral: GLB-SCI — Participants will take part in a lifestyle intervention program (tailored for spinal cord injury needs) that encourages steady weight loss through increased physical activity and healthier diet patterns.
  Arms: GLB-SCI
Behavioral: GLB-SCI+ — Participants will receive a combination of the prior interventions studied, with the goal of showing that a multi-component intervention will be the most effective in encouraging weight loss among participants with a spinal cord injury.
  Arms: GLB-SCI+

SUMMARY:
This study's overarching aim is to follow a systematic approach that incorporates community-based participatory research (CBPR) to develop a multi-component weight loss intervention that may yield significant effects for a chronic SCI sample. The approach is to obtain data on the 3 unique strategies (prepackaged/portion-controlled meals; enhanced self-monitoring; the GLB-SCI) to inform design of an empirically supported and consumer-validated multicomponent intervention program, that combines the best of the 3 approaches into one unique intervention, the GLB SCI+. Based on the investigators' prior experience with adapting and delivering the GLB AIM (a lifestyle intervention previously adapted for those with impaired mobility), interim findings, existing literature, and consumer feedback, they hypothesize that these 3 unique strategies may confer individualized benefits to people with SCI given their complex disability-related barriers to weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Have had a spinal cord injury for at least 1 year
* Overweight as evidenced by BMI > 25
* Must have sufficient upper arm mobility to engage in exercise
* Must have access to the internet
* Must be able to obtain physician signed clearance to participate in a weight management intervention

Exclusion Criteria:

* Cognitive impairment which substantially impairs autonomy (e.g. mental retardation)
* Medical issues for which exercise is contraindicated such as uncontrolled hypertension or coronary heart disease,
* Pregnancy
* Not fluent in English
* Presence of grade 3 or 4 pressure ulcer
* Previously diagnosed eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change in weight | Approximately every 13 weeks through study completion, expected to be 3 years.
  Change in weight (pounds) will be measured after each 13-week intervention.
Change in physical activity level | Approximately every 13 weeks through study completion, expected to be 3 years.
  Change in self-reported physical activity (minutes per week) will be measured after each 13-week intervention to assess whether the intervention effectively encouraged greater levels of physical activity.
Self-efficacy | Approximately every 13 weeks through study completion, expected to be 3 years.
  Self-efficacy will be measured through changes in the Self-Rated Abilities for Health Practices Scale from baseline to post-intervention. The questionnaire contains 28 items that are on a 5-point scale. It was designed to measure a person's perception of his/her own ability to practice "healthy" behaviors and has 4 sub-scales with 7 items each: Exercise, Nutrition, Responsible Health Practice, and Psychological Well Being. Ratings for each subscale are summed to yield subscale scores and subscale scores are summed to obtain a total score. Higher scores indicate greater confidence in one's ability to perform health practices and total scores range from 0-112.
Function/Quality of Life | Approximately every 13 weeks through study completion, expected to be 3 years.
  Changes in self-reported levels of function and quality of life will be assessed through the LIFE-H survey, given before and after each intervention. The Assessment of Life Habits (LIFE-H) assesses a person's self-reported difficulty with and need for assistance performing tasks associated with activities of daily living (ADL) and social roles. The version used for this study covers 6 ADL categories: nutrition, fitness, personal care, communication, residence, mobility and 6 social role categories: responsibility, interpersonal relations, community, education, employment, recreation. Scoring is based on respondent rating of level of accomplishment (No difficulty to Not accomplished) combined with the type of assistance (if any) used to perform these tasks. Scores range from 9 to 0, with higher scores indicating less difficulty.

SECONDARY OUTCOMES:
Change in waist circumference | Approximately every 13 weeks through study completion, expected to be 3 years.
  Participants will have their waist circumference measured before and after each intervention to assess the level of change, if any.
Change in blood pressure (systolic and diastolic) | Approximately every 13 weeks through study completion, expected to be 3 years.
  Participants will have their blood pressure measured before and after each intervention to assess the level of change, if any.
Change in hemoglobin A1c level | Approximately every 13 weeks through study completion, expected to be 3 years.
  Participants will have their hemoglobin A1c measured before and after each intervention assess the level of change, if any.
Change in motivation for weight-loss | Approximately every 13 weeks through study completion, expected to be 3 years.
  Participants will have their levels of motivation assessed before and after each intervention with the Treatment Self-Regulation Questionnaire. The 18-item Treatment Self-Regulation Questionnaire is derived from self-determination theory and yields 2 subscales: autonomous regulation (or intrinsic motivation) and controlled regulation (or extrinsic motivation). Responses are provided on a 7-point Likert type scale ranging from 1 'not at all true' to 7 'very true,' and includes the option of "not applicable." Autonomous Regulation scores are obtained by averaging questions 3, 4, 9, 13, 17, 18 and Controlled Regulation scores are obtained by averaging questions 1, 2, 5, 6, 7, 8, 10, 11, 12, 14, 15, 16. Higher scores indicate higher levels of motivation. Higher scores indicate higher levels of each type of regulation.

OTHER OUTCOMES:
Group meeting attendance | Attendance will be tracked over the entire 13-week intervention.
  Intervention arms involving meeting on a regular basis will have attendance tracked to assess the overall feasibility of the intervention and to examine correlations between self-monitoring and weight-loss.
Adherence to self-monitoring | Adherence will be tracked over the entire 13-week intervention.
  Intervention arms involving self-monitoring food intake and physical activity will have levels of adherence tracked to assess the overall feasibility of the intervention and to examine correlations between self-monitoring and weight-loss.
Individualized teleconference attendance | Attendance will be tracked over the entire 13-week intervention.
  Intervention arms involving teleconference meeting attendance will have levels of adherence tracked to examine correlations between attendance and weight-loss.
Participant perceptions of each intervention | Perception will be assessed at the end of the 13-week intervention.
  Participant perceptions will be assessed using a survey that asks participants to rate on a scale of 1 - 5 each active component used in each study

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Institute for Rehabilitation - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate data designed to study the feasibility, effectiveness, and usability of several weight-loss strategies in a sample of approximately 100 participants with spinal cord injury. These data will be submitted to Inter-university Consortium for Political and Social Research (ICPSR). ICPSR will make the research data from this project available to the broader social science research community. These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, may be accessed directly through the ICPSR website. After depositing the data, the dissemination will be delayed for one year to allow for the principal investigator and collaborators to complete major manuscripts related to the data. ICPSR will accept responsibility for long-term preservation of the research data upon receipt of a signed deposit form.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after completion of all study activities. The research data from this project will be deposited with the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR) to ensure that the research community has long-term access to the data.